CLINICAL TRIAL: NCT01340001
Title: Effects of Nucleus Basalis of Meynert Area Electrical Stimulation on Cognitive Behavioral Disorders in Dementia With Lewy Bodies : A Pilot Phase 1 Study
Brief Title: Effects of Nucleus Basalis of Meynert Stimulation on Cognitive Disorders in Dementia With Lewy Bodies
Acronym: DEMENSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/049/HP; 2011-A00387-34 (Other: ID-RCB)
Record Dates: First submitted 2011-04-05; First posted 2011-04-21 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Dementia With Lewy Bodies
Keywords: Dementia with Lewy bodies; Nucleus basalis of Meynert; Deep brain stimulation
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Electrical stimulation of the nucleus basalis of Meynert (Sham Comparator): Deep brain stimulation
  Interventions: Procedure: Electrical stimulation of the nucleus basalis of Meynert
- Electrical stimulation of the nucleus basalis of Meynert (Experimental): Deep brain stimulation
  Interventions: Procedure: Electrical stimulation of the nucleus basalis of Meynert

INTERVENTIONS:
Procedure: Electrical stimulation of the nucleus basalis of Meynert — Differents parameters will be assessed.

SUMMARY:
Deep brain stimulation has been developed as a substitute for the classical lesioning methods previously used in stereotactic and functional neurosurgery. Recent, anecdotal cases reports suggested that electrical stimulation of the cholinergic output of the Nucleus Basalis of Meynert (NBM) may improve cognitive performances, especially the memory tasks.

The present study aims to assess the effect of bilateral electrical stimulation of the NBM on the mnesic performance [assessed by the sum of the three free recalls of the Free and Cued Selective Recall Reminding Test (FCSRT)] in patients diagnosed with probable, moderate, Dementia with Lewy Bodies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Lewy-body dementia according to the internationally accepted consensus criteria (McKeith, 2005)
* Outpatients, male or female, aged between 18 to 75 years
* Moderate dementia defined by a mini-mental state examination (MMSE) score between 16 and 26
* Stable dose of cholinesterase inhibitors (maximal dose tolerated) for a minimum of 1 months
* Patients receiving antiparkinsonian treatment unmodified for 3 months, if treated
* French as native language
* Written informed consent of the patient
* Written informed consent of the caregiver

Exclusion Criteria:

* Other causes of dementia (Alzheimer dementia, vascular dementia, dementia associated with Parkinson's disease)
* Other causes of extrapyramidal symptoms (Parkinson's disease)
* Patients with a history of severe psychiatric disorders, such as psychosis. Earlier episodes of depression and/or anxiety without hospitalization are not exclusion criteria
* Contraindications for MR imaging (claustrophobia, metallic foreign bodies, pacemakers, etc)
* MRI evidence of cerebral microbleeds
* Surgical contraindications: especially, hemostatic disorders, severe cortical atrophy
* Patients receiving treatments that may interfere with the cholinergic system: anticholinergics, cholinomimetics.
* Patients receiving neuroleptics
* Patients with a history of alcohol or drug abuse
* Pre-existing structural brain abnormalities (such as tumor, infarction, or intracranial hematoma)
* Previous neurosurgical intervention
* Patients with a progressively fatal disease, or life expectancy £ one year
* Asthma
* Severe visual deficit of ophthalmic origin (such as glaucoma, age related macular degeneration, cataract)
* Fertile women not using adequate contraceptive methods
* Women who are pregnant or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10-24 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
free recalls of the FCSRT | between the assessments (Month 7) and (Month 10)
  The primary endpoint of the study is the difference in the sum of the three free recalls of the FCSRT between the assessments (M7) and (M10), i.e. the comparison of the performances with and without NBM electrical stimulation.

SECONDARY OUTCOMES:
performances on different tests | different tests recorded at Month 7 and Month 10
  Comparison will be made between the performances on different tests recorded at M7 and M10, to evaluate the effect of bilateral electrical stimulation of the NBM on cognitivo-behavioral disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GODEFROY, Md, PhD, Principal Investigator — University Hospital of Amiens; Luc DEFEBVRE, MD, PhD, Principal Investigator — University Hospital of Lille; HOUETO Jean-Luc, MD, PhD, Principal Investigator — University Hospital of Poitiers; Pierre Krystkowiak, MD, PhD, Principal Investigator — University Hospital of Amiens; Vincent Delasayette, MD, Principal Investigator — University Hospital of Caen
Locations (1):
- Maltête David, Rouen, France

REFERENCES:
- [Derived] Maltete D, Wallon D, Bourilhon J, Lefaucheur R, Danaila T, Thobois S, Defebvre L, Dujardin K, Houeto JL, Godefroy O, Krystkowiak P, Martinaud O, Gillibert A, Chastan M, Vera P, Hannequin D, Welter ML, Derrey S. Nucleus Basalis of Meynert Stimulation for Lewy Body Dementia: A Phase I Randomized Clinical Trial. Neurology. 2021 Feb 2;96(5):e684-e697. doi: 10.1212/WNL.0000000000011227. Epub 2020 Nov 16. PMID 33199437